CLINICAL TRIAL: NCT02399735
Title: Safety Study of Nature Killer Cells From Sibship to Treat the Recurrence of Hepatocellular Carcinoma After Liver Transplantation
Brief Title: Safety Study of NK Cells From Sibship to Treat the Recurrence of HCC After Liver Transplantation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Wang Guoying, Department of liver transplantation, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: (2014)2-126
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: NK cells; Liver Transplantation; Hepatocellular Carcinoma Recurrence
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A (Experimental): Received conventional treatment and NK cells once per two-week for the first two-month, at a dose of 5×10E9 NK cells.
  Interventions: Biological: Low Dose NK cells ×4 times
- Arm B (Experimental): Received conventional treatment and NK cells once per two-week for the first two-month, at a dose of 1×10E10 NK cells.
  Interventions: Biological: Normal Dose NK cells ×4 times
- Arm C (Experimental): Received conventional treatment and NK cells once per two-week for the first four-month, at a dose of 1×10E10 NK cells.
  Interventions: Biological: Normal Dose NK cells ×8 times

INTERVENTIONS:
Biological: Low Dose NK cells ×4 times — Received conventional treatment and NK cells once per two-week for the first two-month, at a dose of 5×10E9 NK cells.
  Other Names: low dose Natural killer cells ×4 times
  Arms: Arm A
Biological: Normal Dose NK cells ×4 times — Received conventional treatment and NK cells once per two-week for the first two-month, at a dose of 1×10E10 NK cells.
  Other Names: normal dose Natural killer cells ×4 times
  Arms: Arm B
Biological: Normal Dose NK cells ×8 times — Received conventional treatment and NK cells once per two-week for the first four-month, at a dose of 1×10E10 NK cells.
  Other Names: normal dose Natural killer cells ×8 times
  Arms: Arm C

SUMMARY:
The purpose of this study is to explore the safety of NK cells from Sibship in patients with recurrent hepatocellular carcinoma after liver transplantation.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is one of the indications for the liver transplantation. With the advancement of liver transplantation associated science and technology, the recurrence of tumor posttransplantation has become the principal contradiction to worsen the prognosis and therefore the prevention of recurrence of HCC is the key to improve the efficacy of liver transplantation. Adoptive cellular immunotherapy has been applied in various malignant tumors including HCC and has obtained significant effects. But for patients with liver transplant in immunosuppressed states, to successfully apply the immune cells to prevent and treat HCC relapse after liver transplantation must balance immunosuppression and anti-tumor immunity. It is necessary to consider the safety of adoptive cellular immunotherapy,and it is also necessary to consider the effectiveness of treatment that the immune cells in the immunosuppression state can exert anti-tumor effects. Natural killer cells (NK cells) have MHC-unrestricted killing effect on malignant tumor cells and are not major mediating cells for GVHD, and might be an optimum choice to meet the above requirements.

Patients with confirmed recurrence of hepatocellular carcinoma after liver transplantation at the Third Affiliated Hospital of Sun Yat-sen University were enrolled.Participants in the study will be assigned to one of three treatment arms:

Arm A: Participants will received conventional treatment and low dose of NK cells treatment for 4 times. Arm B: Participants will received conventional treatment and normal dose of NK cells treatment for 4 times. Arm C: Participants will received conventional treatment and normal dose of NK cells treatment for 8 times. The cultured NK cells from the peripheral blood of the same blood type were taken and infused at intervals of two weeks. Periodic liver function recheck and imaging examination were conducted for 6 months after the last NK cells infusion.

ELIGIBILITY:
Inclusion Criteria:

* Proved hepatocellular carcinoma histologically after liver transplantation.
* Confirmed recurrence of hepatocellular carcinoma by CT/MRI.
* The same blood type relatives with blood transmitted diseases negative.
* Written informed consent.

Exclusion Criteria:

* Autoimmune diseases require long-term of glucocorticoid.
* Other candidates who are judged to be not applicable to this study by investigators.
* Poor compliance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2014-10; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
GVHD | 6 months
  Rash, fever, diarrhea, jaundice etc. leukocyte, platelet, red blood cells reduce, abnormal liver function.Pathological biopsy if necessary.

SECONDARY OUTCOMES:
Acute rejection | 6 months
  abnormal liver function，pathological biopsy if necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yang, MD, Study Chair — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Wang Guoying, Guangzhou, Guangdong, China